CLINICAL TRIAL: NCT00562315
Title: 18F-FACBC PET-CT for the Detection and Staging of Recurrent Prostate Carcinoma (CA129356-01).
Brief Title: FACBC PET/CT for Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David M. Schuster, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, David M. Schuster, MD, Sponsor-Investigator, Emory University
Organization: Emory University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00006468; R01CA129356-01 (NIH)
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FACBC PET-CT and ProstaScint CT (Other): Participants diagnosed with localized prostate carcinoma with subsequent definitive therapy or suspicion of recurrent cancer will undergo an FACBC PET-CT scan and the ProstaScinct CT.
  Interventions: Drug: FACBC; Other: ProstaScinct

INTERVENTIONS:
Drug: FACBC — Anti-3-[18F]FACBC is an investigational positron emission tomography (PET) radiotracer being studies given intravenously prior to PET scan
  Other Names: Fluciclovine
Other: ProstaScinct — ProstaScint (In-Capromab Pendetide) is used to image the extent of prostate cancer in standard practice. Capromab is a mouse monoclonal antibody which recognizes prostate specific membrane antigen from prostate cancer cells and normal prostate tissue. It is given intravenously prior to undergoing CT imaging.
  Other Names: In-Capromab Pendetide

SUMMARY:
Hypothesis:Anti-[18F]FACBC PET-CT will adequately detect local and extraprostatic recurrence, and lead to better characterization of disease status in restaging patients.

This is a study that will test a compound (chemical substance) that has a small amount of radioactivity attached to it. This substance has a natural tendency to go to prostate tissue. The substance is called [18]FACBC and it is given in the form of an injection into a vein. After the substance reaches the prostate, scans called PET or Positron Emission Tomography, are done. This is similar to having CAT scans or x-rays. Usually a compound called [18]FDG is used for PET scans but this substance is eliminated by the kidneys and cannot reach the prostate. This substance called [18]FACBC is not eliminated by the kidneys and may allow tumors in the prostate to be seen better. It is sometimes difficult to tell if a growth on the prostate is cancer with scans or x-rays that are usually done.

Anti-[18F]FACBC PET-CT will be compared to ProstaScint (In-capromab pendetide) which is the conventional imaging for prostate cancer. Investigators will be blinded of the intervention.

This study will look at how the [18]FACBC goes into the prostate tissue and determine its ability to detect recurrent prostate cancer.

ELIGIBILITY:
STUDY NOW CLOSED for recruitment

Inclusion Criteria:

* Patients must be 18 years of age or older.
* Patients will have been originally diagnosed with localized (Stage T1c, T2, or T3 ) prostate carcinoma and have undergone what was considered definitive therapy for localized disease.
* In the case of brachytherapy, cryotherapy, or external beam radiation, treatment will have occurred at least 2 years in the past to eliminate patients with so-called "PSA bump."
* Patient will have suspicion of recurrent prostate carcinoma as defined by: ASTRO criteria of three consecutive rises of PSA or earlier if clinically appropriate, and/or nadir + 2.0 after radiotherapy, and/or greater than 0.3 after prostatectomy.
* Ability to lie still for PET scanning
* Patients must be able to provide written informed consent.

Exclusion Criteria:

* Age less than 18.
* Greater than T3 disease in past
* Prior prostatectomy or 2 years since brachytherapy, cryotherapy, or external beam radiation therapy.
* Does not meet above criteria of suspicious PSA elevation
* Inability to lie still for PET scanning
* Cannot provide written informed consent.
* Bone scan findings characteristic for metastatic prostate carcinoma
* Less than 2 months since any prior prostate biopsy (to decrease false positive uptake from inflammation).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2007-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Schuster, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Schuster DM, Nieh PT, Jani AB, Amzat R, Bowman FD, Halkar RK, Master VA, Nye JA, Odewole OA, Osunkoya AO, Savir-Baruch B, Alaei-Taleghani P, Goodman MM. Anti-3-[(18)F]FACBC positron emission tomography-computerized tomography and (111)In-capromab pendetide single photon emission computerized tomography-computerized tomography for recurrent prostate carcinoma: results of a prospective clinical trial. J Urol. 2014 May;191(5):1446-53. doi: 10.1016/j.juro.2013.10.065. Epub 2013 Oct 19. PMID 24144687
- [Background] Schuster DM, Savir-Baruch B, Nieh PT, Master VA, Halkar RK, Rossi PJ, Lewis MM, Nye JA, Yu W, Bowman FD, Goodman MM. Detection of recurrent prostate carcinoma with anti-1-amino-3-18F-fluorocyclobutane-1-carboxylic acid PET/CT and 111In-capromab pendetide SPECT/CT. Radiology. 2011 Jun;259(3):852-61. doi: 10.1148/radiol.11102023. Epub 2011 Apr 14. PMID 21493787
- [Background] Amzat R, Taleghani P, Savir-Baruch B, Nieh PT, Master VA, Halkar RK, Lewis MM, Faurot M, Bellamy LM, Goodman MM, Schuster DM. Unusual presentations of metastatic prostate carcinoma as detected by anti-3 F-18 FACBC PET/CT. Clin Nucl Med. 2011 Sep;36(9):800-2. doi: 10.1097/RLU.0b013e318219b47e. PMID 21825855
- [Background] Jani AB, Fox TH, Whitaker D, Schuster DM. Case study of anti-1-amino-3-F-18 fluorocyclobutane-1-carboxylic acid (anti-[F-18] FACBC) to guide prostate cancer radiotherapy target design. Clin Nucl Med. 2009 May;34(5):279-84. doi: 10.1097/RLU.0b013e31819e51e3. PMID 19387202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was completed November 28,2007 through July 10, 2012.
Pre-assignment Details: Of the 128 participants consented, 93 participants met the criteria to receive the ProstaScint (In-capromab pendetide) and the FACBC (anti-3-[18F]) scans. 115 participants had FACBC scans, with 13 receiving repeat scans. Therefore, excluding 13 participants. 93 participants had one FACBC scan and one ProstaScint scan and did not have repeat scans.
Groups:
- FACBC PET-CT and ProstaScint CT: Participants diagnosed with localized prostate carcinoma with subsequent definitive therapy or suspicion of recurrent cancer underwent an FACBC PET-CT scan and the ProstaScinct CT.
Period: Overall Study
Arm/Group | FACBC PET-CT and ProstaScint CT
Started | 93
Completed | 93
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants completed both the FACBC PET-CT and the ProstaScint CT.
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 93
Region of Enrollment [Number; unit: participants]
  United States | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With True Positive Scans Within the Prostate Bed
Description: Total number of participants with positive FACBC PET-CT and ProstaScint CT scans in diagnosis of prostate cancer in the prostate bed validated by prostate biopsy and follow up.
Time Frame: Up to 5 years
Population: 91 participants had sufficient data to determine disease presence or absence in the prostate bed.
Measure: Number; unit: participants
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 91
participants
  FACBC PET-CT | 55
  ProstaScint CT | 41

2. Primary Outcome: Number of Participants With False Positive Scans Within the Prostate Bed
Description: Total number of participants with positive FACBC PET-CT and ProstaScint scans in the prostate bed that were confirmed as negative by biopsy and or follow up.
Time Frame: Up to 5 years
Population: 91 participants had sufficient data to determine disease presence or absence in the prostate bed.
Measure: Number; unit: participants
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 91
participants
  FACBC PET-CT | 18
  ProstaScint CT | 13

3. Primary Outcome: Number of Participants With True Negative Scans Within the Prostate Bed
Description: Total number of participants with negative FACBC PET-CT and ProstaScint CT scans in the prostate bed that were confirmed as negative by biopsy and or follow up.
Time Frame: Up to 5 years
Population: 91 participants had sufficient data to determine disease presence or absence in the prostate bed.
Measure: Number; unit: participants
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 91
participants
  FACBC PET-CT | 12
  ProstaScint CT | 17

4. Primary Outcome: Number of Participants With False Negative Scans Within the Prostate Bed
Description: Total number of participants with negative FACBC PET-CT and ProstaScint CT scans in the prostate bed that were confirmed as positive by biopsy and or follow up.
Time Frame: Up to 5 years
Population: 91 participants had sufficient data to determine disease presence or absence in the prostate bed.
Measure: Number; unit: participants
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 91
participants
  FACBC PET-CT | 6
  ProstaScint CT | 20

5. Primary Outcome: Number of Participants With True Positive Scans Outside the Prostate Bed
Description: Total number of participants with positive FACBC PET-CT and ProstaScint CT scans outside the prostate bed (extra-prostate) that were confirmed as positive by biopsy and/or follow up.
Time Frame: Up to 5 years
Population: There was sufficient data for 70 participants to determine disease presence or absence at extraprostatic locations.
Measure: Number; unit: participants
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 70
participants
  FACBC PET-CT | 22
  ProstaScint CT | 4

6. Primary Outcome: Number of Participants With True Negative Scans Outside the Prostate Bed
Description: Total number of participants with negative FACBC PET-CT and ProstaScint CT scans outside the prostate bed (extra-prostate) that were confirmed as negative by biopsy and/or follow up.
Time Frame: Up to 5 years
Population: There was sufficient data for 70 participants to determine disease presence or absence at extraprostatic locations.
Measure: Number; unit: participants
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 70
participants
  FACBC PET-CT | 29
  ProstaScint CT | 26

7. Primary Outcome: Number of Participants With False Positive Scans Outside the Prostate Bed
Description: Total number of participants with positive FACBC PET-CT and ProstaScint CT scans outside the prostate bed (extra-prostate) that were confirmed as negative by biopsy and/or follow up.
Time Frame: Up to 5 years
Population: There was sufficient data for 70 participants to determine disease presence or absence at extraprostatic locations.
Measure: Number; unit: participants
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 70
participants
  FACBC PET-CT | 1
  ProstaScint CT | 4

8. Primary Outcome: Number of Participants With False Negative Scans Outside the Prostate Bed
Description: Total number of participants with negative FACBC PET-CT and ProstaScint CT scans outside the prostate bed (extra-prostate) that were confirmed as positive by biopsy and/or follow up.
Time Frame: Up to 5 years
Population: There was sufficient data for 70 participants to determine disease presence or absence at extraprostatic locations.
Measure: Number; unit: participants
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 70
participants
  FACBC PET-CT | 18
  ProstaScint CT | 36

9. Primary Outcome: Diagnostic Performance of Anti-[18F]FACBC PET-CT Imaging in Detection of Extra-prostatic Recurrence of Prostate Carcinoma
Description: 1. Sensitivity = How well FACBC PET is able to correctly detect when there is prostate cancer outside the prostate bed. [total number of true positives / total number of study participants confirmed to have prostate cancer outside the prostate bed (True positives + False negatives)]
  2. Specificity = How well FACBC PET is able to correctly detect when there is no prostate cancer outside the prostate bed. [ total number of true negatives / total number of study participants confirmed to not have prostate cancer outside the prostate bed (True negatives + False positives)]
  3. Accuracy = (True positives + true negatives)/all tests
  4. Positive predictive value = probability that subjects with a positive screening test truly have prostate cancer outside the prostate bed
  5. Negative predictive value = probability that subjects with a negative screening test truly don't have prostate cancer outside the prostate bed
Time Frame: Up to 5 years
Population: Participants with a definitive consensus for the presence or absence of extraprostatic disease.
Measure: Number (95% Confidence Interval); unit: percentage of true tests
Groups:
- FACBC PET/CT for Recurrent Prostate Cancer: This is a single arm study
  [18F]FACBC: [18F]FACBC is given intravenously prior to PET scan
Arm/Group | FACBC PET/CT for Recurrent Prostate Cancer
Number analyzed (Participants) | 70
percentage of true tests
  % Sensitivity | 55.0 [38.5 to 70.7]
  % Specificity | 96.7 [82.8 to 99.9]
  % Accuracy | 72.9 [60.9 to 82.8]
  % Positive Predictive Value | 95.7 [78.1 to 99.9]
  % Negative Predictive Value | 61.7 [46.4 to 75.5]

10. Primary Outcome: Diagnostic Performance of Anti-[18F]FACBC PET-CT Imaging in Detection of Recurrent Prostate Carcinoma in the Prostate Bed
Description: 1. Sensitivity = How well FACBC PET is able to correctly detect when there is prostate cancer in the prostate bed. i.e. total number of true positives / total number of study participants confirmed to have prostate disease in the prostate bed (True positives + False negatives)
  2. Specificity = How well FACBC PET is able to correctly detect when there is no prostate cancer in the prostate bed. i.e. total number of true negatives / total number of study participants confirmed to not have prostate disease in the prostate bed (True negatives + False positives)
  3. Accuracy = (True positives + true negatives)/all tests
  4. Positive predictive value = the probability that subjects with a positive screening test truly have prostate carcinoma in the prostate bed
  5. Negative predictive value = the probability that subjects with a negative screening test truly don't have prostate carcinoma in the prostate bed
Time Frame: Up to 5 years
Population: Participants with a definitive consensus on the presence or absence of prostatic/bed disease.
Measure: Number (95% Confidence Interval); unit: percentage of true tests
Groups:
- FACBC PET/CT for Recurrent Prostate Cancer: Participants diagnosed with localized prostate carcinoma with subsequent definitive therapy or suspicion of recurrent cancer underwent an FACBC PET-CT scan and the ProstaScinct CT.
Arm/Group | FACBC PET/CT for Recurrent Prostate Cancer
Number analyzed (Participants) | 91
percentage of true tests
  % Sensitivity | 90.2 [79.8 to 96.3]
  % Specificity | 40.0 [22.7 to 59.4]
  % Accuracy | 73.6 [63.3 to 82.3]
  % Positive Predictive Value | 75.3 [63.9 to 84.7]
  % Negative Predictive Value | 66.7 [41.0 to 86.7]

11. Secondary Outcome: Diagnostic Performance of ProstaScint Imaging in Detection of Recurrent Prostate Carcinoma in the Prostate Bed
Description: 1. Sensitivity = How well ProstaScint imaging is able to correctly detect when there is prostate cancer in the prostate bed. i.e. total number of true positives / total number of study participants confirmed to have prostate disease in the prostate bed (True positives + False negatives)
  2. Specificity = How well ProstaScint imaging is able to correctly detect when there is no prostate cancer in the prostate bed. i.e. total number of true negatives / total number of study participants confirmed to not have prostate disease in the prostate bed (True negatives + False positives)
  3. Accuracy = (True positives + true negatives)/all tests
  4. Positive predictive value = the probability that subjects with a positive screening test truly have prostate carcinoma in the prostate bed
  5. Negative predictive value = the probability that subjects with a negative screening test truly don't have prostate carcinoma in the prostate bed
Time Frame: Up to 5 years
Population: Participants with a definitive consensus on the presence or absence of prostatic/bed disease.
Measure: Number (95% Confidence Interval); unit: percentage of true tests
Arm/Group | FACBC PET/CT for Recurrent Prostate Cancer
Number analyzed (Participants) | 91
percentage of true tests
  % Sensitivity | 67.2 [54.0 to 78.7]
  % Specificity | 56.7 [37.4 to 74.5]
  % Accuracy | 63.7 [53.0 to 73.6]
  % Positive Predictive Value | 75.9 [62.4 to 86.5]
  % Negative Predictive Value | 45.9 [29.5 to 63.1]

12. Secondary Outcome: Diagnostic Performance of ProstaScint Imaging in Detection of Extra-prostatic Recurrence of Prostate Carcinoma
Description: 1. Sensitivity = How well ProstaScint is able to correctly detect when there is prostate cancer outside the prostate bed. [total number of true positives / total number of study participants confirmed to have prostate cancer outside the prostate bed (True positives + False negatives)]
  2. Specificity = How well ProstaScint is able to correctly detect when there is no prostate cancer outside the prostate bed. [ total number of true negatives / total number of study participants confirmed to not have prostate cancer outside the prostate bed (True negatives + False positives)]
  3. Accuracy = (True positives + true negatives)/all tests
  4. Positive predictive value = the probability that subjects with a positive screening test truly have prostate cancer outside the prostate bed
  5. Negative predictive value is the probability that subjects with a negative screening test truly don't have prostate cancer outside the prostate bed
Time Frame: Up to 5 years
Population: Participants with a definitive consensus for the presence or absence of extraprostatic disease.
Measure: Number (95% Confidence Interval); unit: percentage of true tests
Arm/Group | FACBC PET-CT and ProstaScint CT
Number analyzed (Participants) | 70
percentage of true tests
  % Sensitivity | 10.0 [2.8 to 23.7]
  % Specificity | 86.7 [69.3 to 96.2]
  % Accuracy | 42.9 [31.1 to 55.3]
  % Positive Predictive Value | 50.0 [15.7 to 84.3]
  % Negative Predictive Value | 41.9 [29.5 to 55.2]

ADVERSE EVENTS:
Groups:
- FACBC PET-CT and ProstaScint CT: All participants who received scans, including repeat scans, were monitored for adverse events.
Arm/Group | FACBC PET-CT and ProstaScint CT
Serious Adverse Events (participants affected / at risk) | 0/115
Other Adverse Events (participants affected / at risk) | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No